CLINICAL TRIAL: NCT00551785
Title: The Multinational Postmarketing Observational Study of Women Prescribed Intrinsa
Brief Title: Surveillance Study of Women Taking Intrinsa®
Acronym: EMPOWER
Status: Terminated | Type: Observational
Why Stopped: The marketing authorization for Intrinsa was withdrawn.
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Principal Investigator, Klaas Heinemann, MD, PhD, Principal Investigator, Center for Epidemiology and Health Research, Germany
Other Study IDs: ZEG2007_01
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Ovariectomy; Hysterectomy; Hypoactive Sexual Desire Disorder
Keywords: Hypoactive Sexual Desire Disorder; Menopause; Androgen
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Women prescribed Intrinsa and estrogen therapy
- 2: Women prescribed estrogen therapy

SUMMARY:
The primary objective of the study is to assess the risks of testosterone transdermal patch use in a representative study population. The primary clinical outcome of interest is breast cancer.

DETAILED DESCRIPTION:
This is a prospective, controlled, non-interventional long-term cohort study of women who are prescribed estrogen therapy or estrogen therapy in combination with Intrinsa®.

Intrinsa® is a transdermal patch that delivers 300 mcg of testosterone daily through the skin of the abdomen, providing women with testosterone levels that are within the physiological range for premenopausal women. It is indicated for the treatment of hypoactive sexual desire disorder (HSDD) in women with bilateral oophorectomy and hysterectomy who are receiving concomitant estrogen therapy.

A non-interference approach will be used to provide standardized, comprehensive, reliable information on these treatments under routine medical conditions.

The two main objectives of this study are:

* to estimate the incidence of breast cancer, other gynecological cancer, myocardial infarction, other cardiovascular outcomes and other rare serious adverse outcomes among Intrinsa® users in actual clinical practice, and
* to compare these incidences with the incidences found in the comparison group of women with bilateral oophorectomy and hysterectomy using estrogen therapy.

The primary variable for the statistical analysis is the breast cancer hazard ratio for Intrinsa® users in comparison to users of estrogen therapy.

The secondary objectives of the study are:

* to analyze the Intrinsa® utilization pattern in a study population that is representative for the users of this novel treatment
* to characterize the baseline risk of Intrinsa® users for breast cancer and cardiovascular diseases and
* to investigate the reversibility of specific androgenic outcomes after stop of treatment.

The two study cohorts will consist of new users of Intrinsa® in combination with estrogen therapy and estrogen therapy without simultaneous use of Intrinsa®, respectively. After study entry cohort members will be followed for a period of five to eight years for rare serious safety outcomes. Regular, active contacts with the cohort members by the ZEG study team (=active surveillance) will provide the necessary information on health-related events or changes in health status. All cohort members will be contacted at 6 and 12 months after study entry, and then every 12 months.

Approximately 5.400 subjects per cohort will be recruited by participating physicians in order to provide 50.000 women-years (WY) of observation, assuming a withdrawal rate of 10% per year. Enrollment procedures should not interfere with the prescribing behavior of physicians or with the individual needs of the participating women.

The study will be conducted in Italy, France, Spain, the UK and Germany. It could be extended to other countries based on the international registration and launch status of Intrinsa®.

The study will be divided into two phases: a clinic phase, which includes an initial consultation at baseline with a participating physician, and a follow-up phase, which includes two follow-up contacts within the first year, and then annual follow-up contacts for up to eight years post-baseline.

The study participants are women who have a new prescription of Intrinsa® in combination with estrogen therapy or estrogen therapy respectively and who are willing to participate in this cohort study. There are no specific medical inclusion or exclusion criteria other than the guidance provided by the local product label. However, women who are not cooperative may be excluded from study participation. Also women with a language barrier will not be eligible for study inclusion.

This study will maintain scientific independence and will be governed by an independent Advisory Council. The Center for Epidemiology and Health Research in Berlin, Germany and its research team will be accountable for the Advisory Council (AC) in all scientific matters. The members of the AC wil be international experts in relevant scientific fields (e. g. epidemiology, gynecology and cardiology).

Information on the identity of the patients and treating physicians will be kept separated from the clinical information throughout the study. All relevant national data protection laws will be followed.

ELIGIBILITY:
Inclusion Criteria:

* All women with bilateral oophorectomy and hysterectomy who receive a new prescription for the study medication or who were prescribed it for a period of six months or less before study entry

Exclusion Criteria:

* Women who at baseline have used Intrinsa® or the new estrogen therapy for more than six months
* Women who do not consent to participate in the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women prescribed estrogen therapy or estrogen therapy in combination with Intrinsa
Sampling Method: Non-Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2007-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
gynecological cancer; serious cardiovascular diseases | Time to event analysis within 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Klaas Heinemann, MD, PhD, Principal Investigator — Center for Epidemiology and Health Research, Germany
Locations (1):
- Center for Epidemiology and Health Research, Berlin, Germany